CLINICAL TRIAL: NCT07375758
Title: A Phase I/II, Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of MIL116 in Healthy Participants and Patients With IgA Nephropathy
Brief Title: A Study of MIL116 in Healthy Participants and Patients With IgA Nephropathy.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Mabworks Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIL116-CT101
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Immunoglobulin A Nephropathy
Keywords: Anti-APRIL monoclonal antibody; MIL116; IgAN
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIL116 (Experimental)
  Interventions: Drug: MIL116
- Placebo (Placebo Comparator)
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: MIL116 — MIL116 is supplied as sterile solution for subcutaneous (SC) injection.
  Arms: MIL116
Drug: Matching Placebo — Placebo is to be administered at a matching volume by SC injection.
  Arms: Placebo

SUMMARY:
This is a Phase I/II study designed to evaluate the safety, tolerability, PK and PD of subcutaneous MIL116, an anti-APRIL monoclonal antibody, in healthy participants and patients with IgA Nephropathy.

ELIGIBILITY:
Inclusion Criteria:

-

Phase Ia:

1. Able to understand and voluntarily sign the written Informed Consent Form (ICF), willing and able to comply with all study requirements;
2. Healthy participants aged 18 to 55 years (inclusive) at the time of signing the ICF, of either sex;
3. Have a body mass index (BMI) between 19 to 32 kg/m² (inclusive) and a body weight ≥ 50 kg at screening;
4. Assessed to be in good health status based on medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests, with no clinically significant abnormalities;
5. Have a total immunoglobulin G (IgG) level > 10 g/L at screening; and immunoglobulin A (IgA) and immunoglobulin M (IgM) levels within the normal reference ranges.

Phase Ib&II:

1. Able to understand and voluntarily sign the written ICF, and willing and able to comply with all study requirements;
2. Aged ≥ 18 years at the time of signing the ICF, of either sex, with a BMI ≥ 16 kg/m²;
3. Biopsy-confirmed diagnosis of IgA Nephropathy (IgAN). Participants must have a 24-hour urine protein-to-creatinine ratio (UPCR) ≥ 0.5 g/g or 24-hour urine protein ≥ 0.75 g prior to the first dose;
4. Have been receiving an optimized and stable dose of an angiotensin-converting enzyme inhibitor (ACEi) or angiotensin II receptor antagonist (ARB). If currently receiving sodium-glucose cotransporter 2 inhibitors (SGLT2i) and / or endothelin receptor antagonists (ERA), the same administration and dose stability requirements apply for;
5. Have acceptable hematologic, hepatic, coagulation, and renal function as assessed by clinical laboratory tests.

Exclusion Criteria:

-

Phase Ia:

1. Nursing, lactating or pregnant, or who have plans to become pregnant during the study
2. History or evidence of any clinically significant disease, disorder, or condition that, in the investigator's judgment, may pose a risk to the participants' safety, interfere with the study assessments, or render the subject unsuitable for participation, including but not limited to respiratory, renal, hepatic, gastrointestinal, hematological, lymphatic, neurologic, cardiovascular, psychiatric, or other systemic diseases;
3. Any confirmed or suspected immunosuppressive or immunodeficiency condition, including human immunodeficiency virus (HIV) infection or asplenia; history of recurrent or severe infections, or long-term use of immunosuppressive agents within 6 months prior to screening;
4. History of chronic infection (e.g., tuberculosis, osteomyelitis) or any infectious disease requiring hospitalization or treatment with antiviral, antibiotic, or antifungal agents within 28 days prior to administration of the study drug;
5. Use of any prescription medications, over-the-counter (OTC) drugs, herbal products, topical products, or dietary supplements within 28 days prior to administration of the study drug or for within 5 half-lives of the drug (whichever is longer);
6. Participation in any clinical study of an investigational drug or medical device, or receipt of any investigational study drug, within 3 months prior to administration of the study drug or within 5 half-lives (whichever is longer);
7. Receipt of any marketed or investigational antibody or biologic therapy (including immunoglobulin products, monoclonal antibodies, or antibody fragments) within 28 days prior to administration of the study drug or within 5 half-lives (whichever is longer);
8. History of drug abuse or substance dependence, or a positive urine drug abuse screening result during the screening period.

Phase Ib&II:

1. Secondary IgAN or IgA vasculitis (Henoch-Schönlein purpura), as diagnosed by the investigator;
2. Presence of chronic kidney disease of causes other than IgAN;
3. Other significant pathological abnormalities identified on kidney biopsy;
4. Kidney biopsy demonstrating tubular-interstitial fibrosis > 50% or glomerular crescents involving > 25% of glomeruli. Note: The most recent kidney biopsy will be prioritized for eligibility assessment;
5. Clinical suspicion of rapidly progressive glomerulonephritis based on an estimated glomerular filtration rate (eGFR) decline ≥ 50% within 3 months prior to the screening visit;
6. Nephrotic syndrome, defined as 24-hour urine protein > 3.5 g accompanied by hypoalbuminemia (serum albumin < 30 g/L). Subjects with isolated nephrotic-range proteinuria (> 3.5 g/d) are excluded;
7. Receipt of rituximab or any B-cell depleting agent within 6 months prior to screening. Participants with CD4+ T-cell count < 200 cells/μL are excluded;
8. Total IgG level < 6 g/L at screening; uncontrolled type 2 diabetes mellitus, defined as glycated hemoglobin (HbA1c) > 8%; or diagnosis of type 1 diabetes mellitus;
9. History of prior treatment with any APRIL-targeted medication;
10. Receipt of biologic agents, such as belimumab or eculizumab, within 3 months prior to the first dose of the study drug;
11. Receipt of cyclophosphamide within 3 months prior to the first dose; use of other immunosuppressive agents within 28 days prior to the first dose, including but not limited to azathioprine, mycophenolate mofetil, leflunomide, tacrolimus, cyclosporine, methotrexate, or tripterygium wilfordii; systemic corticosteroids used at an average daily dose equivalent to ≥40 mg prednisone for more than 14 days within 28 days prior to the screening visit, or use of oral delayed-release budesonide capsules within 1 year prior to the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Safety and Tolerability of Single Ascending Doses of MIL116 in Healthy Participants. | up to 6 months after enrollment
  Percentage of Participants with AEs and SAEs assessed by NCI CTCAE v5.0.
Phase Ib: Safety and Tolerability of Multiple-Ascending Doses of MIL116 in IgAN Participants. | up to 18 months after enrollment
  Description: Percentage of Participants with AEs and SAEs assessed by NCI CTCAE v5.0.
Phase II: Change in Gd-IgA1 from Baseline at Week 12 | up to 18 months after enrollment
  Evaluate the degree and percentage change of Gd-IgA1 from baseline.
Change in 24-Hour Urine UPCR from Baseline at Week 24 | up to 18 months after enrollment
  Evaluate the degree and percentage change of 24-hour urine UPCR from baseline